CLINICAL TRIAL: NCT04020549
Title: Evaluating the Effectiveness of a Computerized, School-Based, Single-Session Intervention for Rural Indian Adolescents
Brief Title: Single-Session Computerized Mental Health Intervention for Rural Indian Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: In collaboration with community partners, we determined that the reading level required for the intervention did not make it suitable for the adolescents.
Sponsor: University of Pennsylvania (Other)
Collaborators: Sangath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 30927492
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Well-Being; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Growth

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Growth, Gratitude, & Positive Activities
- Study Skills Control (Sham Comparator)
  Interventions: Behavioral: Study Skills Control

INTERVENTIONS:
Behavioral: Growth, Gratitude, & Positive Activities — Reading and writing activities based on growth (designed to instill the belief that people can change), gratitude (noticing and appreciating good things in life), and behavioral activation (identifying and scheduling positive activities).
  Arms: Intervention
Behavioral: Study Skills Control — Reading and writing activities designed to teach evidence-based study strategies.
  Arms: Study Skills Control

SUMMARY:
The overall aim of this project is to understand if single-session interventions are acceptable, culturally appropriate, and effective for Indian adolescents attending a rural, low-resource government school. The investigators will be examining the effects of a computerized intervention on the well-being and mental health of adolescents. The investigators hypothesize that the intervention will yield statistically significant improvements in wellbeing and mental health relative to a study skills control condition.

ELIGIBILITY:
Inclusion Criteria:

* Attending a participating secondary school
* Age 12 to 18
* Literate in English

Exclusion Criteria:

* Unable to provide informed consent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in The Warwick-Edinburgh Mental Wellbeing Scale | Baseline, 4 week follow-up, 12 week follow-up
  Well-being questionnaire. Total score ranges from 14 to 70. Higher values indicate a better outcome.
Intervention Appropriateness Measure | Immediately post-intervention (i.e., 0 weeks)
  Questionnaire measuring the appropriateness of an intervention. Appropriateness refers to the perceived fit or relevance of an intervention. The total score ranges from 4 to 20. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Baseline, 4 week follow-up, 12 week follow-up
  Depression Questionnaire. The total score ranges from 0 to 27. Lower scores indicate a better outcome.
Generalized Anxiety Disorder Screener-7 | Baseline, 4 week follow-up, 12 week follow-up
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
The EPOCH Measure of Adolescent Well-being | Baseline, 4 week follow-up, 12 week follow-up
  Questionnaire with five subscales measuring engagement, perseverance, optimism, connectedness, and happiness. Each subscale score ranges from 4 to 20. Higher scores indicate a better outcome. The happiness and optimism subscales will be used as secondary outcomes for this trial. A total score is not computed.
Acceptability of Intervention Measure | Immediately post-intervention (i.e., 0 weeks)
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Feasibility of Intervention Measure | Immediately post-intervention (i.e., 0 weeks)
  Questionnaire measuring the feasibility of an intervention. Feasibility refers to the degree to which a treatment can be successfully implemented in a given setting. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Perceived Stress Scale-4 | Time Frame: Baseline, 4 week follow-up, 12 week follow-up
  Questionnaire measuring perceived stress. The total score ranges from 0 to 16. Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rob DeRubeis, PhD, Study Director — University of Pennsylvania; Sachin Shinde, PhD, Study Director — Sangath; Sadhana Natu, PhD, Study Director — Modern College Pune; Akash Wasil, Principal Investigator — University of Pennsylvania
Locations (1):
- Z P school, Wablewadi, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No